CLINICAL TRIAL: NCT03715608
Title: Total Knee Arthroplasty Combined With Psychological Intervention for Patients With Psychological Disorders to Improve Postoperative Outcome and Patient Satisfaction
Brief Title: Total Knee Arthroplasty Combined With Psychological Intervention for Patients With Psychological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Tian Hua, vice director of department of orthopaedics, Peking University Third Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tianhua68480
Record Dates: First submitted 2018-10-14; First posted 2018-10-23 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee; Psychological Disorder; Psychological Intervention; Satisfaction; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Mental Disorders; Personal Satisfaction | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the control group received routine TKA surgery and perioperative management without any other interventions.
- Intervention group (Experimental): The patients in the intervention group received professional psychological interventions include psychological counseling and corresponding medication after the operation. Other perioperative treatments were the same as the patients in the control group. Psychotherapy was based on the clinical expertise of the psychosocial specialist, who selected the most appropriate plan for each patient.
  Interventions: Other: Psychological Intervention

INTERVENTIONS:
Other: Psychological Intervention — The patients in the intervention group received psychological counseling and corresponding medication after the operation. Psychotherapy was based on the clinical expertise of the psychosocial specialist from Peking University Sixth Hospital, who selected the most appropriate plan for each patient.
  Arms: Intervention group

SUMMARY:
Objective To evaluate the incidence of psychological problems in total knee arthroplasty (TKA) patients and examine whether perioperative psychological intervention can improve the outcomes of and patient satisfaction with TKA.

Methods The investigators will prospectively collect clinical data from 400 patients who underwent primary TKA by the same surgeon at Peking University Third Hospital. The patients will be divided into 3 groups based on psychological status and intervention: the normal group comprised patients with a normal psychological status, while patients with an abnormal psychological status will be randomly divided into the intervention group, which received psychological interventions, and the control group, which do not receive any psychological interventions. The HSS（Hospital of special surgery） and WOMAC scores will be evaluated preoperatively, 3 months postoperatively and 6 months postoperatively. A self-administered satisfaction scale (very satisfied, somewhat satisfied, somewhat dissatisfied, very dissatisfied) that assessed overall satisfaction as well as satisfaction with pain relief and the ability to perform daily and leisure activities will be administered 6 months postoperatively.

Hypothesis A certain percentage of TKA patients have preoperative psychological abnormalities. Preoperative psychological abnormalities can have an adverse effect on postoperative improvement in joint function and can reduce patient satisfaction. Preoperative psychological intervention can improve the prognosis of TKA patients with psychological disorders.

DETAILED DESCRIPTION:
Patients with knee osteoarthritis（OA） undergoing primary unilateral TKA at the Department of Orthopedics of Peking University Third Hospital from May 2016 to January 2018 will be prospectively included in the study. Inclusion criteria: (1) Signed written informed consent; (2) Willingness to complete the assessment and an examination using a psychometric scale; (3) No surgical contraindications. Exclusion criteria: (1) Patients undergoing revision; (2) Patients with infection; (3) Patients who could not undergo the psychological assessment; (4) Loss to follow-up; (5) Psychological disorders of severe type, which means the patient needs to stop TKA surgery for psychological therapy. The patients' general preoperative data and joint function scores will be collected. Preoperative psychoanalysis will be conducted by a psychiatrist from Peking University Sixth Hospital to determine the TKA patients' preoperative psychological characteristics.

According to the presence or absence of psychological abnormalities, the patients will be divided into a psychological abnormalities group and a normal group. The patients in the normal group will receive routine TKA surgery and perioperative management without any other interventions.

A randomized controlled prospective study will be conducted with the patients in the psychological abnormalities group. They will be randomly divided into two groups: the intervention group and the control group.

The control group: Like the patients in the normal group, the patients in the control group will receive routine TKA surgery and perioperative management without any other interventions.

The intervention group: The patients in the intervention group will receive psychological counseling and corresponding medication after the operation. Other perioperative treatments will be the same as the patients in the control group. Psychotherapy will be based on the clinical expertise of the psychosocial specialist, who will select the most appropriate plan for each patient.

The WOMAC and HSS scores of all patients will be analyzed preoperatively, 3 months postoperatively and 6 months postoperatively, and a postoperative satisfaction survey questionnaire will be completed.

For every patient in this study, standard TKA and perioperative management will be performed by one experienced surgeon at Peking University Third Hospital. Postoperative follow-up will be performed by a group of doctors who are blinded to the group and intervention information.

Psychological status assessment and clinical outcome evaluation The patients' psychological and physical performance will be assessed using the Symptom Checklist (SCL-90), a self-assessment questionnaire that is commonly used to assess patients' psychological health. The SCL-90 has a good ability to identify people with psychological symptoms (especially patients on the border of clinically significant psychological symptoms).

To assess whether a patient had a psychological disorder that met the diagnostic criteria before surgery, the MINI-International Neuropsychiatric Interview (MINI) will be used to assess patients with suspected anxiety or depression. The MINI is a short, structured interview for the diagnosis of Diagnostic and Statistical Manual-IV（DSM-IV）and International Classification of Diseases-10（ICD-10 ） axis psychiatric disorders. It can be conducted in a short period of time (average 15 minutes). The Chinese version of the MINI has shown reliability and validity in clinical practice. It has been widely used clinically in China.

The HSS and WOMAC scores will be evaluated preoperatively, 3 months postoperatively and 6 months postoperatively.

A self-administered satisfaction scale (very satisfied, somewhat satisfied, somewhat dissatisfied, very dissatisfied) that assessed overall satisfaction as well as satisfaction with pain relief and the ability to perform daily and leisure activities will be administered 6 months postoperatively.

Psychological intervention There are three main interventions for TKA patients: patient visits and education, medication, and psychological interventions.

1. Patient visits and education: Patient education can shorten hospital stays, reduce surgical complications, relieve preoperative anxiety and depressive symptoms, increase confidence, and improve patient satisfaction. In particular, patients with clear psychological problems should pay attention to and divert disease-related negative emotions, such as tension, fear, depression and anxiety.
2. Drug treatment：Patients who meet the indications for drug treatment should be treated with drugs that are sensitive and effective as recommended by psychiatrists.

   2.1 Antidepressants are usually divided into tricyclic antidepressants, tetracyclic antidepressants, monoamine oxidase inhibitors, selective serotonin reuptake inhibitors (SSRIs), dopamine reuptake inhibitors, serotonin and desmethyl selective serotonin and norepinephrine reuptake inhibitors (SNRIs), norepinephrine and specific serotonin antidepressants. Among them, SSRIs and SNRIs are widely used in clinical practice. The SSRIs are fluoxetine hydrochloride, paroxetine hydrochloride, sertraline, fluvoxamine, citalopram and escitalopram. The main SNRI drugs are venlafaxine, duloxetine and milnacipran.

   2.2 Anti-anxiety drugs are mainly benzodiazepines, such as diazepam, alprazolam, and clonazepam, and aromatic piperazine anxiolytics, such as buspirone.
3. Psychological interventions include cognitive and behavioral therapy, supportive therapy, relaxation therapy, and such methods as group therapy, motivational interview therapy, and interpersonal psychotherapy.

Each patient has his or her own psychological characteristics. It most effective for a psychiatrist to develop a personalized psychological intervention program based on the patient's psychological characteristics.

Ethics approval This study has been approved by the Ethics Committee of Peking University Third Hospital. The enrolled patients can choose to withdraw unconditionally at any time during the study, and the investigators guarantee that the patient's TKA surgery would continue unaffected.

Statistical analysis The data distribution will be normal according to the Kolmogorov-Smirnov test. Descriptive statistics will be used to analyze the demographic data and other baseline features, and the number, mean, and standard deviation values will be calculated for continuous variables. Pearson correlations and paired T tests for preoperative and postoperative data comparisons will be used to evaluate the relationship between different variables. The inferential statistics results (P values) are listed as descriptive results. SPSS (Version 19, SPSS, Inc., Chicago IL) will be used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Willingness to complete the assessment and an examination using a psychometric scale
* No surgical contraindications.

Exclusion Criteria:

* Patients undergoing revision;
* Patients with infection;
* Patients who could not undergo the psychological assessment;
* Loss to follow-up;
* Psychological disorders of severe type, which means the patient needs to stop TKA surgery for psychological therapy.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with TKA surgery Satisfaction | 6 months
  A self-administered satisfaction scale (very satisfied, somewhat satisfied, somewhat dissatisfied, very dissatisfied) that assessed overall satisfaction as well as satisfaction with pain relief and the ability to perform daily and leisure activities was administered 6 months postoperatively.

SECONDARY OUTCOMES:
HSS(Hospital for Special Surgery) score | 6 months
  HSS(hospital for special surgery) score HSS(hospital for special surgery) score to evaluate patients postoperative knee joint function. With a total of 100, it has 7 subscales: 1.Pain 0~30; 2. Function 0~22; 3. Mobility 0~18; 4. Flexion deformity 0~10; 6. Stability 0~10; 7. Deduction Item. For each scale, a higher value represents a better outcome. The sum of the subscales is the total score.
WOMAC(The western Ontario and McMaster universities osteoarthritis index) score | 6 months
  WOMAC(The western Ontario and McMaster universities osteoarthritis index) score HSS(hospital for special surgery) score to evaluate patients postoperative knee joint function.